CLINICAL TRIAL: NCT03976934
Title: Prophylactic Administration of Alpha Blockers for Prevention of Post Operative Urinary Retention in Males Undergoing Open Inguinal Hernia Repair Under Spinal Anaesthesia.
Brief Title: Prophylactic Administration of Alpha Blockers for Prevention of Urinary Retention in Males Undergoing Inguinal Hernia Repair Under Spinal Anaesthesia.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgios Koukoulis (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Sponsor-Investigator, Georgios Koukoulis, General Surgery Consultant, General Hospital of Larissa
Organization: General Hospital of Larissa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1725
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Inguinal Hernia; Urinary Retention
Keywords: open inguinal hernia repair; spinal anaesthesia; urinary retention; elective alpha blockers
MeSH Terms: conditions — Hernia, Inguinal; Urinary Retention | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamsulosin group (Active Comparator): administration of 0,4mg of tamsulosin 24 hours before surgery and 0,4mg 6 hours before surgery
  Interventions: Drug: Tamsulosin
- Placebo group (Placebo Comparator): administration of placebo 24 and 6 hours before surgery
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Tamsulosin — administration of tamsulosin tablets
  Other Names: omnic tocas
  Arms: Tamsulosin group
Drug: Placebo oral tablet — sugar pills
  Arms: Placebo group

SUMMARY:
Open inguinal hernia repair is one of the most common surgical procedures. Despite the fact that different of anesthetic procedures are proposed as alternatives to spinal anesthesia, the combination of spinal anesthesia with open inguinal hernia repair is preferred from both surgeons and patients. One disadvantage of this combination is the high incidence of post-surgery urinary retention, especially in men above 50 years old. This complication is partially attribute to overstimulation of the a1 adrenergic receivers of the bladder and the prostate. Preoperative administration of elective a1 blockers could inhibit this effect without side effects, since this drugs don't have systemic effect.

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia

Exclusion Criteria:

* ASA score >3
* hypotension
* prostatic hypertrophy
* complicated inguinal hernia
* neurological diseases
* inguinal hernia repair under general or local anaesthesia

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
incidence of urinary retention | 8 hours post surgery
  inability to voluntarily void urine up to 8 hours post surgery

SECONDARY OUTCOMES:
Prostate related Symptoms | Baseline
  identification of Prostate related Symptoms as preoperative risk factor of post surgery urinary retention. For the assessment of the prostate related symptomatology will be used the International Prostate Symptom Score questionnaire
Scrotal hernia Repair | Baseline, Inta-operative
  evaluation of Scrotal hernia repair as preoperative risk factor of post surgery urinary retention.
Duration of Surgery | Duration of Surgical procedure
  Evaluation of the surgery duration as inta-operative risk factor of post surgery urinary retention.
Use of opioids | 24 hours
  Evaluation of the peri-operative administration of iv opioids as a peri-operative risk factor of post surgery urinary retention.
Iv fluid administration | 24 hours
  Evaluation of the peri-operative iv fluid administration as a peri-operative risk factor of post surgery urinary retention.
Post-operative Pain | 24 hours
  Evaluation of the post operative pain as a risk factor of post surgery urinary retention. For the assessment of the pain will be used the Visual Analog Scale (VAS) score at 6, 12 and 24 hours after surgery. (VAS Score Scale from 0-10, 0 no pain, 10 max pain)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tepetes, MD, PHD, Study Chair — University Hospital of Larisa and Medical School, University of Thessaly; Georgios D Koukoulis, MD, PhD, Principal Investigator — General Hospital of Larissa; Konstantinos Mpouliaris, MD, Principal Investigator — General Hospital of Larissa
Locations (2):
- Greece (2):
  - University General Hospital of Larissa, Larissa
  - General Hospital Of Larissa, Larissa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clancy C, Coffey JC, O'Riordain MG, Burke JP. A meta-analysis of the efficacy of prophylactic alpha-blockade for the prevention of urinary retention following primary unilateral inguinal hernia repair. Am J Surg. 2018 Aug;216(2):337-341. doi: 10.1016/j.amjsurg.2017.02.017. Epub 2017 Mar 14. PMID 28341140
- [Background] Basheer A, Alsaidi M, Schultz L, Chedid M, Abdulhak M, Seyfried D. Preventive effect of tamsulosin on postoperative urinary retention in neurosurgical patients. Surg Neurol Int. 2017 May 10;8:75. doi: 10.4103/sni.sni_5_17. eCollection 2017. PMID 28584678
- [Background] Shaw MK, Pahari H. The role of peri-operative use of alpha-blocker in preventing lower urinary tract symptoms in high risk patients of urinary retention undergoing inguinal hernia repair in males above 50 years. J Indian Med Assoc. 2014 Jan;112(1):13-4, 16. PMID 25935942